CLINICAL TRIAL: NCT04197141
Title: Is Hypofractionated Whole-Pelvis Radiotherapy (WPRT) as Well Tolerated as Conventionally-Fractionated WPRT in Prostate Cancer Patients? (HOPE-Trial)
Brief Title: Hypofractionated Whole-Pelvis Radiotherapy (WPRT) vs Conventionally-Fractionated WPRT in Prostate Cancer
Acronym: HOPE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Association of Radiation Oncology (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOPE Trial
Record Dates: First submitted 2019-12-06; First posted 2019-12-12 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
Keywords: Unfavorable intermediate risk; High risk
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventionally-fractionated WPRT (Active Comparator): 15 Gy HDR brachytherapy boost will be administered followed by 45 Gy WPRT in 25 fractions. Androgen Deprivation Therapy (ADT) may also be prescribed at the discretion of the treating physician.
  Interventions: Radiation: Conventionally-fractionated WPRT
- Hypofractionated WPRT (Experimental): 15 Gy HDR brachytherapy boost will be administered followed by 25 Gy WPRT in 5 fractions. Androgen Deprivation Therapy (ADT) may also be prescribed at the discretion of the treating physician.
  Interventions: Radiation: Hypofractionated WPRT

INTERVENTIONS:
Radiation: Conventionally-fractionated WPRT — Total dose: 45 Gy in 25 fractions WPRT
  Arms: Conventionally-fractionated WPRT
Radiation: Hypofractionated WPRT — Total dose: 25 Gy in 5 fractions WPRT
  Arms: Hypofractionated WPRT

SUMMARY:
The purpose of this research study is to determine if 5 (five) fractions of external radiotherapy with higher radiation doses per fraction to the pelvis leads to similar results to the standard of care external radiotherapy treatment that is comprised of 25 fractions of external radiotherapy with lower radiation doses per fraction to the pelvis.

This study aims to investigate the impact in quality of life associated with hypofractionated Whole Pelvis Radiotherapy (WPRT) in comparison to conventionally-fractionated WPRT in patients with unfavorable-intermediate and high-risk prostate cancers. This information is valuable as hypofractionated WPRT is a more attractive and convenient treatment approach, and may become the new standard of care if proven to be well-tolerated and effective. Therefore, this study aims to provide a more rational justification for use of hypofractionated WPRT in future larger randomized trials by comparing this strategy with the current standard of care. This study will also provide an initial understanding of the toxicity profile and cancer control associated with hypofractionated WPRT and High Dose Rate Brachytherapy (HDR-BT).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Study Informed Consent provided
* Pathologically proven diagnosis of prostatic adenocarcinoma
* Unfavorable intermediate risk [with greater than 15% chance of node involvement based on Memorial Sloan Kettering Cancer Center (MSKCC) nomogram https://www.mskcc.org/nomograms/prostate] or high or very-high-risk prostate cancer based on National Comprehensive Cancer Network (NCCN) classification [Prostatic Specific Antigen (PSA) > 20 ng/mL or clinical cT3a or cT3b or Gleason 8-10]
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* No prior history of pelvic irradiation, brachytherapy, cryosurgery, High-Intensity Focused Ultrasound (HIFU), Transurethral Resection of the Prostate (TURP) or radical prostatectomy

Exclusion Criteria:

* Presence of nodal or distant metastasis, as confirmed by Magnetic Resonance Imaging (MRI) or Computerized Tomography (CT) of the chest/abdomen/pelvis and bone scan within 45 days of randomization
* Plan for adjuvant docetaxel post-radiotherapy
* Serious medical comorbidities or other contraindications to HDR-BT
* Presence of inflammatory bowel disease
* Presence of connective tissue disease
* Medically unfit for general anesthesia
* Unable or unwilling to complete questionnaires

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QOL) - late bowel function as measured by the EPIC questionnaire | I year post treatment (approximately 3 years and 2 months)
  Late bowel function as reported by the patient using the standardized questionnaire Expanded Prostate Cancer Index Composite (EPIC) sub-domain approximately 1 year after the end of treatment. The EPIC questionnaire contains 32 questions measuring patient function. Each question has a response option ranging from 0 or 1 (best) to 3, 4, or 5 (worst). The responses then correlate to a scoring scale of 0 to 100, where 0 is the best and 100 is the worst. The values vary from 0 to 100 for each question. The scores can then be added to come up with an overall quality of life score.

SECONDARY OUTCOMES:
Quality of Life - acute urinary and sexual QOL as measured by the EPIC questionnaire | 6 weeks post treatment (approximately 2 years and 3 months)
  Acute urinary and sexual QOL as reported by the patient using the standardized questionnaire Expanded Prostate Cancer Index Composite (EPIC) urinary and sexual domains. The EPIC questionnaire contains 32 questions measuring patient function. Each question has a response option ranging from 0 or 1 (best) to 3, 4, or 5 (worst). The responses then correlate to a scoring scale of 0 to 100, where 0 is the best and 100 is the worst. The values vary from 0 to 100 for each question. The scores can then be added to come up with an overall quality of life score.
Quality of Life - acute bowel toxicity as measured by the EPIC questionnaire | 6 weeks post treatment (approximately 2 years and 3 months)
  Acute bowel function as reported by the patient using the standardized questionnaire Expanded Prostate Cancer Index Composite (EPIC) approximately 6 weeks after the end of treatment. The EPIC questionnaire contains 32 questions measuring patient function. Each question has a response option ranging from 0 or 1 (best) to 3, 4, or 5 (worst). The responses then correlate to a scoring scale of 0 to 100, where 0 is the best and 100 is the worst. The values vary from 0 to 100 for each question. The scores can then be added to come up with an overall quality of life score.
Quality of Life - late bowel bother as measured by the EPIC questionnaire | I year post treatment (approximately 3 years and 2 months)
  Late bowel bother as reported by the patient using the standardized questionnaire Expanded Prostate Cancer Index Composite (EPIC) sub-domain approximately 1 year after the end of treatment. The EPIC questionnaire contains 32 questions measuring patient function. Each question has a response option ranging from 0 or 1 (best) to 3, 4, or 5 (worst). The responses then correlate to a scoring scale of 0 to 100, where 0 is the best and 100 is the worst. The values vary from 0 to 100 for each question. The scores can then be added to come up with an overall quality of life score.
Quality of Life - late urinary and sexual QOL as measured by the EPIC questionnaire | I year post treatment (approximately 3 years and 2 months)
  Late urinary and sexual QOL as reported by the patient using the standardized questionnaire Expanded Prostate Cancer Index Composite (EPIC). The EPIC questionnaire contains 32 questions measuring patient function. Each question has a response option ranging from 0 or 1 (best) to 3, 4, or 5 (worst). The responses then correlate to a scoring scale of 0 to 100, where 0 is the best and 100 is the worst. The values vary from 0 to 100 for each question. The scores can then be added to come up with an overall quality of life score.
International Prostate Symptom Score (IPSS) | 6 weeks post treatment (approximately 2 years and 3 months), 1 year post treatment (approximately 3 years and 2 months) and 2 years post treatment (approximately 4 years and 2 months)
  International Prostate Symptom Score (IPSS) as reported by the patient at 6 weeks, 1 year, and 2 years post treatment. The IPSS is a tool used for monitoring symptoms of prostate enlargement (benign prostatic hyperplasia). There are 7 questions related to urinary function. Responses are on a scale from 0 (best) to 5 (worst). Responses are added to come up with a total score, measuring if the patient is mildly symptomatic, moderately symptomatic, or severely symptomatic. There is 1 quality of life question related to urinary symptoms. Responses are on a scale from 0 (best) to 6 (worst).
Toxicity - urinary, bowel, and sexual as measured by CTCAE version 4.0 | 6 weeks post treatment (approximately 2 years and 3 months), 1 year post treatment (approximately 3 years and 2 months) and 2 years post treatment (approximately 4 years and 2 months)
  Urinary, bowel, and sexual toxicity will be measured by the Common Terminology Criteria for Adverse Events (CTCAE) version 4, at 6 weeks, 1 year, and 2 years post treatment.
Prostatic Specific Antigen (PSA) curve | 4 years post treatment (approximately 6 years and 2 months)
  PSA curve at 4 years post-treatment.
Prostatic Specific Antigen (PSA) Nadir | 4 years post treatment (approximately 6 years and 2 months)
  PSA nadir at 4 years post-treatment.
Cost Effectiveness of Hypofractionated WPRT | End of study (approximately 7 years and 2 months)
  Cost effectiveness analysis of the hypofractionated arm in comparison to the conventionally fractionated treatment arm.
Overall Survival | End of study (approximately 7 years and 2 months)
  The time from randomization to death from any cause.
Biochemical Failure-Free Survival | End of study (approximately 7 years and 2 months)
  The time from randomization to biochemical failure (based on the Phoenix definition) or death from any cause, whichever occurs first.
Freedom from Local Failure | End of study (approximately 7 years and 2 months)
  The time from randomization to first local failure.
Freedom from Regional Failure | End of study (approximately 7 years and 2 months)
  The time from randomization to first regional failure.
Androgen Deprivation Therapy Free Survival | End of study (approximately 7 years and 2 months)
  The time from randomization to start of salvage ADT, death or last follow-up.
Metastasis Free Survival | End of study (approximately 7 years and 2 months)
  The time from randomization to development of metastasis, death or last follow-up.
Prostate Cancer Free Survival | End of study (approximately 7 years and 2 months)
  The time from randomization to death attributed to prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas C Mendez, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (3):
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BC Cancer, Kelowna, British Columbia
  - London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mendez LC, Arifin AJ, Bauman GS, Velker VM, Ahmad B, Lock M, Venkatesan VM, Sexton TL, Rodrigues GB, Chen J, Schaly B, Warner A, D'Souza DP. Is hypofractionated whole pelvis radiotherapy (WPRT) as well tolerated as conventionally fractionated WPRT in prostate cancer patients? The HOPE trial. BMC Cancer. 2020 Oct 9;20(1):978. doi: 10.1186/s12885-020-07490-0. PMID 33036579